CLINICAL TRIAL: NCT06526910
Title: Your Mind Can Exercise Too: A Novel Application of Motor Imagery Practice in Swallowing Rehabilitation
Brief Title: Your Mind Can Exercise Too: Swallowing Motor Imagery Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samford University (Other)
Collaborators: Case Western Reserve University (Other); Emerson College (Other); James Madison University (Other); Texas Christian University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: EXPD-HP-24-S-6
Record Dates: First submitted 2024-07-02; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This is a multiple baselines single case series study. Each participant will complete 4 sequential phases of the study. Phase 1 is standard of care dysphagia exercise (baseline), Phase 2 is wash-out (no exercise, Phase 3 is standard of care + motor imagery practice OR continued standard of care exercise only, and Phase 3 is a second wash-out period (no exercise).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 Standard of Care (Active Comparator): A four-week period of standard of care dysphagia treatment consisting of physical swallowing-related exercises. According to guidelines for single case design, this standard of care treatment will serve as a baseline/control period for comparison to the subsequent experimental treatment period. Participants will complete either 6, 7, or 8 baseline measurement visits across these 4 weeks (multiple baseline design).
  Interventions: Behavioral: Swallowing exercises
- Phase 2 Wash-out period #1 (No Intervention): A three-week wash-out period. All participants will attend 6 measurement sessions across the 3-week period but will not complete any swallowing exercises.
- Phase 3 "Experimental" (Experimental): A four-week exercise period. Five participants will be assigned to complete a second period of standard of care swallowing exercises while the other five will be assigned to the experimental treatment which includes standard of care plus motor imagery practice. According to single case design, participants will complete either 6, 7, or 8 measurement visits across these 4 weeks.
  Interventions: Behavioral: Swallowing exercises
- Phase 4 Wash-out period #2 (No Intervention): A final three-week wash-out period. All participants will attend 6 measurement sessions across the 3-week period but will not complete either the standard of care or the experimental swallowing exercises.

INTERVENTIONS:
Behavioral: Swallowing exercises — Standard-of-care swallowing exercises include tongue exercise. The experimental part added in Phase 3 includes some participants completed standard-of-care exercises again and others completing standard-of-care exercises and motor imagery practice of those exercises.
  Arms: Phase 1 Standard of Care; Phase 3 "Experimental"

SUMMARY:
Swallowing difficulty (dysphagia) is a clinical symptom of Parkinson's disease (PD) that significantly impacts nutrition, oral secretion management, health status, and quality of life]. Specific hallmarks of dysphagia in patients with PD include tongue weakness, reduced swallowing frequency and efficiency, and airway invasion. Evidence for effective treatment techniques to address dysphagia in patients with PD is limited and urgently needed, substantiating the systematic study of standard-of-care treatments in this population as well as the development of novel techniques. Motor imagery practice (MIP) is a mentally rehearsed form of exercise that does not involve muscle activation and has been shown to improve motor outcomes in limb rehabilitation. MIP is novel to swallowing rehabilitation. Our group has conducted preliminary MIP studies in healthy older adults and demonstrated improved measures of tongue strength and swallowing pressure when MIP is used in combination with physical tongue exercise compared to physical tongue exercise alone. The next step is to evaluate the use of MIP in patients with dysphagia. The purpose of this research is to determine the feasibility and effect of MIP when added to a physical swallowing-related exercise protocol for patients with PD. Changes in tongue pressure generation, spontaneous swallowing frequency, functional physiological swallowing outcomes, and patient-reported outcomes will be examined. This research aims to fill gaps in evidence specific to dysphagia in patients with PD and to evaluate a novel rehabilitation method. The investigators anticipate that the results of this study will inform clinical practice, with evidence for supporting the improvement of swallowing function and quality of life in patients with PD, and lay the groundwork for the design of future randomized controlled clinical trials.

DETAILED DESCRIPTION:
The proposed study is a five-site research collaboration between Samford University (Birmingham, AL, Dr. Sarah Szynkiewicz), Case Western Reserve University (Cleveland, OH, Dr. Rachel Mulheren), Emerson College (Boston, MA, Dr. Lindsay Griffin), James Madison University (Harrisonburg, VA, Dr. Erin Kamarunas), and Texas Christian University (Fort Worth, TX, Dr. Teresa Drulia). The Samford IRB serves as the main IRB, with the other sites executing IRB Authorized Agreements with Samford's IRB. The research sessions will be conducted in each site PI's university laboratory and each site PI will be responsible for overseeing the recruitment and data collection at their respective site. Standardized forms and training to both the protocol and data analysis will be completed across all sites and will ensure research fidelity.

The investigators will conduct a multiple baseline single case study (n = 10) to determine feasibility and explore the preliminary effects of motor imagery practice (MIP) on swallowing function in patients with Parkinson's disease (PD). Single case designs are often used as an initial exploration of treatment efficacy prior to a randomized controlled trial. Using this prospective design, participants with PD will complete:

* Phase 1: A four-week period of standard of care dysphagia treatment consisting of physical swallowing-related exercises. According to guidelines for single case design, this standard of care treatment will serve as a baseline/control period for comparison to the subsequent experimental treatment period. Participants will complete either 6, 7, or 8 baseline measurement visits across these 4 weeks (multiple baseline design).
* Phase 2: A three-week wash-out period. All participants will attend 6 measurement sessions across the 3-week period but will not complete any swallowing exercises.
* Phase 3: A four-week exercise period. Five participants will be assigned to complete a second period of standard of care swallowing exercises while the other five will be assigned to the experimental treatment which includes standard of care plus motor imagery practice. According to single case design, participants will complete either 6, 7, or 8 measurement visits across these 4 weeks.
* Phase 4: A final three-week wash-out period. All participants will attend 6 measurement sessions across the 3-week period but will not complete either the standard of care or the experimental swallowing exercises.

The findings of this single case design study will inform the feasibility of methods and provide an estimate of rehabilitation outcomes that will lead to the development of larger randomized controlled clinical trials to determine the efficacy of this promising, novel MIP approach to swallowing rehabilitation in PD and other patient populations with dysphagia. The investigators anticipate this research will confirm the feasibility of using motor imagery practice (MIP) to improve swallowing-related outcomes for patients with Parkinson's disease (PD). The investigators hypothesize that patients with PD will demonstrate a faster rate of improved tongue pressure and spontaneous swallowing frequency during the four-week physical swallowing-related exercise + MIP practice protocol (experimental treatment) compared to the four weeks of physical exercise only (standard of care treatment). Furthermore, the investigators hypothesize that these changes will result in greater improvements in swallowing efficiency and safety (as measured objectively using instrumental swallowing assessment) at the end of treatment. The investigators also expect to provide preliminary evidence that spontaneous swallowing frequency can be used as a measure of functional change in swallowing in patients with PD when instrumental evaluation cannot be accessed or used in repetition.

ELIGIBILITY:
Inclusion criteria. Individuals will be able to participate if they:

* Are >/= 65 years of age as this is an independent predictor for dysphagia in PD
* Are diagnosed with moderate-stage Parkinson's disease (Hoehn & Yahr disease stage 2-3)
* Disease duration >3 years as this in an independent predictor for dysphagia in PD
* Are currently managed using an antiparkinsonian medication, including at least one dopaminergic drug (i.e., carbidopa/levodopa or a dopamine agonist)
* Have reduced tongue strength, defined as < 45 kilopascals when completing a maximal isometric tongue push using the standard IOPI procedures
* Present with some dysphagia symptoms, defined as a score > 3 on the Eating Assessment Tool (EAT-10)
* Have some mental imagery ability, defined as a score > 2.5 greater on the KVIQ-10 short version
* Present with signs of dysphagia that are clinically detectable, as defined by a score < 178 on the Mann Assessment of Swallowing Ability (MASA)
* Are cognitively able to participate, as defined by a score > 19 on the telephone Montreal Cognitive Assessment (T-MoCA)
* Have a normal oral structure as assessed with a standardized oral mechanism exam
* Are fluent in English as all instruction will be provided in English

Exclusion criteria. Individuals will not be eligible to participate if they report:

* Changes to their dopaminergic medication management anytime during enrollment
* They are currently recommended by a Speech-Language Pathologist to have NPO (nothing by mouth) status for safety reasons
* A history of oral surgery (routine dental surgery acceptable)
* Additional neurogenic disorders other than Parkinson's disease
* A history of swallowing difficulty prior to Parkinson's disease diagnosis
* A history of seizures
* A history of cancer that would impact oral-motor function
* A history of allergy to barium
* That they have initiated deep brain stimulation less than 3 months from the start of the study, or that they are anticipated to have a change in deep brain stimulation status during participation in the study
* Participation in other swallowing, speech, or voice treatments outside of the research treatment at the time of consent and anytime during enrollment
* Demonstration of normal swallowing function on first study-related modified barium swallow test, defined as a level 6 or higher on the Dysphagia Outcome and Severity Scale (DOSS). Therefore, participants must get a DOSS of 5 or lower, indicating at least mild oropharyngeal dysphagia, at baseline testing before beginning the treatment protocol. This reduces the risk of a null finding by eliminating the enrollment of participants with functional swallows or subclinical swallowing issues.
* A current pain disorder involving the jaw muscles or joint of the mandible (i.e., TMJ disorder or myofascial pain disorder)
* Not being available to complete a 16-week in-person study protocol
* Known or suspected perforation of the gastrointestinal (GI) tract
* Known obstruction of the GI tract
* High risk of GI perforation such as those with a recent GI perforation, acute GI hemorrhage or ischemia, toxic megacolon, severe ileus, post GI surgery or biopsy, acute GI injury or burn, or recent radiotherapy to the pelvis
* High risk for aspiration such as those with known or suspected tracheo-esophageal fistula or obtundation
* Known hypersensitivity to barium sulfate or any of the excipients of Varibar pudding

No potential participant will be excluded on the basis of race, color, creed, sex, sexual orientation, or national origin.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale score | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  The most severe level of airway invasion will be determined using the Penetration and Aspiration Scale, an eight-point nominal scale (0-8, 8 representing the most severe form of airway invasion) that allows the clinical to define the depth of food/liquid entering the airway and the patient response to it (e.g., coughing).

SECONDARY OUTCOMES:
Tongue pressures | Multiple timepoints across the study as part of the single case series study design, e.g., baseline, up to twice a week during each Phase, post-intervention
  Maximum isometric pressure and regular saliva swallow pressure measures (continuous scale, e.g., 0-100+ kilopascals
Spontaneous swallowing frequency | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  Spontaneous swallowing frequency will be measured using a microphone and digital voice recorder to record swallowing sounds at rest for a 10-minute period. The audio recording will be analyzed off-line. Continuous scale, e.g. 0-10+ swallows/minute
Swallowing-related quality-of-life | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  The participant will complete a self-reported validated swallowing-related quality-of-life questionnaire, The Dysphagia Handicap Index, (25-items with up to 4 points assigned for each question by the participant, 0-100 points, with a higher score indicating a worse quality-of-life rating).
Radboud Oral Motor Inventory for Parkinson's disease (ROMP) | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  The saliva portion of the ROMP will be completed as a validated patient-reported outcome for oral secretion management. The saliva sub-scale is 9 questions with up to 5 points each assigned by the participants, 0-45 points, with a higher score indicating a worse issue managing saliva).
Dysphagia severity level | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  Severity of dysphagia will be determined using the Dysphagia Outcome and Severity Scale, a seven-point ordinal scale allowing the clinician to define the patient's swallowing severity from normal to severely impacted.
Oral transit time | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  Oral transit time (OTT) reflects the duration (in milliseconds) required to move a bolus through the oral cavity and reflects lingual strength and coordination. OTT will be defined as the time interval between the beginning of posterior bolus movement in the oral cavity to when the bolus tail passes the posterior nasal spine indicating the bolus has passed through the oral cavity. Longer oral transit times suggest reduced swallowing efficiency.
Laryngeal vestibule closure (LVC) reaction time | Measured at 3 timepoints across the study for each participant: baseline, immediately after Phase 1 intervention, immediately after Phase 3 intervention
  LVC reaction time reflects the time required for the laryngeal vestibule to close once the swallowing reflex has been initiated. LVC reaction time will be defined as the time interval between when the hyoid has the initial anterior-superior "jump" and the first frame showing contact (or maximum approximation) between the arytenoid process and the inferior surface of the epiglottis. Longer LVC reaction times suggest reduced swallowing safety.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Szynkiewicz, PhD, Principal Investigator — Samford University

IPD SHARING:
Plan to Share IPD: No